CLINICAL TRIAL: NCT03410290
Title: The Journey of Patients With Vasculitis From First Symptom to Diagnosis
Brief Title: Journey of Patients With Vasculitis From First Symptom to Diagnosis
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Peter Merkel, Chief, Division of Rheumatology, Professor of Medicine and Epidemiology, University of Pennsylvania
Other Study IDs: VCRC5538/V-PPRN4
Record Dates: First submitted 2018-01-18; First posted 2018-01-25 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Vasculitis; Systemic Vasculitis; Behcet's Disease; CNS Vasculitis; Cryoglobulinemic Vasculitis; Eosinophilic Granulomatous Vasculitis; Temporal Arteritis; Giant Cell Arteritis; Granulomatosis With Polyangiitis; Wegener Granulomatosis; Henoch Schonlein Purpura; IgA Vasculitis; Microscopic Polyangiitis; Polyarteritis Nodosa; Takayasu Arteritis; Urticarial Vasculitis
MeSH Terms: conditions — Vasculitis; Systemic Vasculitis; Behcet Syndrome; Vasculitis, Central Nervous System; Cryoglobulinemia, Familial Mixed; Churg-Strauss Syndrome; Giant Cell Arteritis; Granulomatosis with Polyangiitis; IgA Vasculitis; Microscopic Polyangiitis; Polyarteritis Nodosa; Takayasu Arteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: The online questionnaire includes questions about factors that impacted a patients diagnosis of vasculitis.
  Interventions: Other: Online Questionnaire

INTERVENTIONS:
Other: Online Questionnaire — The online questionnaire includes questions about factors that impacted a patients diagnosis of vasculitis.

SUMMARY:
This study seeks to understand the journey that patients eventually are diagnosed with vasculitis experience in the period prior to their formal diagnosis by a healthcare provider. Data elements of interest include average time from the onset of the first symptoms to the time a diagnosis of vasculitis is confirmed. Other aims include identifying factors associated with the time to diagnosis. These factors will be divided into: a) intrinsic factors, or so-called "patient-related factors", such as the type of vasculitis symptoms, patient demographics, socioeconomic status, patients' beliefs regarding the etiology of their symptoms, and other factors, and b) extrinsic factors, or "professional/health system factors", such as healthcare access, referral patterns, testing patterns, and other factors. Understanding such factors can guide future efforts to shorten delays in diagnosis and thereby improve outcomes. All analyses will be done for the population of patients with vasculitis as a whole and by individual types of vasculitis.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of a systemic vasculitis: The V-PPRN includes patients with self-reported Behçet's disease, central nervous system vasculitis, cryoglobulinemic vasculitis, eosinophilic granulomatosis with polyangiitis (Churg-Strauss Syndrome, CSS), giant cell (temporal) arteritis (GCA), granulomatosis with polyangiitis (Wegener's, GPA), IgA vasculitis (Henoch-Schönlein Purpura), microscopic polyangiitis (MPA), polyarteritis nodosa (PAN), Takayasu's arteritis (TAK), and urticarial vasculitis.
2. Language requirements: questionnaire will be in English only

Exclusion Criteria:

1. Inability to provide informed consent and complete survey in English
2. Patients with a diagnosis of "other" type of vasculitis
3. Patients with a "missing" diagnosis -

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All individuals with self-reported vasculitis participating in the Vasculitis Patient-Powered Research Network (V-PPRN) will be invited to join the study, with a target recruitment period of 3 months. This study is open to US and international participants.
Sampling Method: Non-Probability Sample
Enrollment: 456 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2018-05-21 (Actual); Study Completion 2018-05-21 (Actual)

PRIMARY OUTCOMES:
Percentages of patients with different types of vasculitis who report a delay in their disease diagnosis from initial symptoms of vasculitis to establishment of a diagnosis of vasculitis, stratified by disease type. | 1 day
  Analysis of how people fill in the questionnaire to determine the time from onset of symptoms of vasculitis to the first encounter with a healthcare provider for evaluation of those symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Sreih, MD, Study Chair — University of Pennsylvania; Peter A Merkel, MD, MPH, Study Director — University of Pennsylvania
Locations (1):
- University of South Florida, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Vasculitis Patient-Powered Research Network — https://www.vpprn.org/